CLINICAL TRIAL: NCT07170748
Title: Clinical Performance Evaluation of MagIA In-vitro Diagnostic Medical Device for Multiplex Screening of Human Immunodeficiency Virus (HIV), Hepatitis B, Hepatitis C and Syphilis in Sub-Saharan Africa
Brief Title: Clinical Performance Evaluation of MagIA IVD-MD Multiplex Testing (HIV/HBV/HCV/Syphilis)
Acronym: MAGICS IBCS
Status: Recruiting | Type: Observational
Sponsor: MagIA Diagnostics (Industry)
Collaborators: Institut Pasteur (Industry); Kenya Medical Research Institute (Other); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other)
Responsible Party: Sponsor
Other Study IDs: MAGIA-H3S-EP-01
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiplex Testing of HIV, HBV, HCV and Syphilis; HIV; HBV; HCV; Syphilis; Point of Care Testing
Keywords: point of care test; HIV; HBV; HCV; Syphilis; multiplex testing
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Performance study to evaluate the clinical performance of the In-Vitro Diagnostics Medical Device MagIA H3S (a Multiplex Point-of-Care test for the combined detection of Human Immunodeficiency Virus (HIV), Hepatitis B and C and Syphilis) from serum, plasma samples collected prospectively or retrospectively in Ivory Coast and Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent for participation in this study.
* Patient sample must meet at least one of the criteria below:

  1. Positive samples (serum or plasma) from individuals who meet at least one of the following conditions:
* HIV-1 Ab positive
* HIV-2 Ab positive
* HCV-Ab positive
* HBsAg positive
* Positive for at least TPHA, with those positive for both TPHA and VDRL ideally included 2. Negative samples (serum or plasma) from individuals who meet at least one of the following conditions:
* Blood donors
* Hospitalized patients or individuals coming to the clinic
* Vulnerable populations (such as: drug users, prison population, ...) 3. Negative samples (serum or plasma) containing potential interfering substances from individuals who meet at least one of the following conditions:
* Being a pregnant woman
* Infected with at least one of the following viruses or bacteria: hepatitis A virus (HAV), hepatitis E virus (HEV), tuberculosis (TB), gonorrhoea, chlamydia, influenza virus, Covid-19
* Presenting any of the following criteria:

  * High IgG levels
  * High rheumatoid factor (>15 IU/mL)
  * High cholesterol levels (>0.24 md/dL)
  * High bilirubin levels (>0.25 mg/mL)
  * High triglyceride levels (>500 mg/dL)
  * Diagnosis of cancer

Exclusion Criteria:

* Samples from patients below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of blood samples from individuals recruited from those seeking viral load testing and diagnostic services for HIV, HBV, HCV, and syphilis or from individuals belonging to one of the target populations of the study
Sampling Method: Non-Probability Sample
Enrollment: 2950 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation of MagIA H3S in detection of HIV-Ab, HBAg, HCV-Ab and TP-Ab | Baseline
  Diagnostic sensitivity (Se), specificity (Sp), positive predictive value (PPV), and negative predictive value (NPV) of the MagIA H3S device for detecting each of the four markers: HIV-Ab, HCV-Ab, HBsAg, and TP-Ab, compared to reference standard testing.

SECONDARY OUTCOMES:
Evaluation of cross-reactivity with any potentially interfering substances or interferences with any co-infection or comorbidity | Baseline
  Identification and collection of suspected and predefined cross-reacting or interfering substances (e.g. alcohol, tobacco, concomitant medication) and comorbidities (e.g. HTLV, EBV, CMV, HSV, malignancy).
  Samples with inconclusive results from MagIA test and those with discordant results between MagIA and reference tests will be further examined for the presence of cross-reacting substances or underlying comorbidities that may influence the signal of the MagIA H3S test. Identified interfering substances will be documented through eCRF and additional analytical investigations will be conducted to confirm their impact.
Evaluation of performance of MagIA H3S in determining on-going HCV infection | Baseline
  Sensitivity, specificity, positive predictive value, and negative predictive value of the MagIA H3S HCV score to detect on-going HCV infection compared to the gold standard, considering only those with positive RNA viral load assay as positive for HCV.

CONTACTS AND LOCATIONS:
Locations (2):
- Centre de Diagnostic et de Recherche sur le SIDA et les autres Maladies Infectieuses - CHU Treichville, Abidjan, Côte d’Ivoire
- Kenya Medical Research Institute (KEMRI), Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No
IPD belonging to the patients are confidential and shall not be shared. It is not planned in the protocol.

REFERENCES:
- See also: Related Info — https://magia-diagnostics.com/project-magfa/